CLINICAL TRIAL: NCT03651973
Title: Prevention of Sequelae Pain After Breast Cancer Surgery by Daily Self Massages and Self Stretching of Serratus Anterior Muscle, Pectoralis Major Muscle, Infraspinatus Muscle and Latissimus Dorsi Muscle: Impact of Learning Workshops Performed by a Multidisciplinary Team.
Brief Title: Prevention of Sequelae Pain After Breast Cancer Surgery by Self-massages and Self Stretching. Impact of Learning Workshops.
Acronym: ESTAUVAL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-4-6-003
Record Dates: First submitted 2018-07-04; First posted 2018-08-29 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Surgery
Keywords: Self massages and self stretching; Workshops for self massages and stretching learning
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With learning workshops (Experimental): Patients in experimental arm will attend learning workshops, one before breast cancer surgey and one after surgery. Patients will be educated by physiologist to self massages and self stretching. Each workshop will last around 2 hours.
  Interventions: Other: Learning workshops
- Without learning workshops (Other): Standard follow-up. Patients randomized in this arm won't attend Learning workshops and will be followed in a standard way.
  Interventions: Other: Standard follow-up

INTERVENTIONS:
Other: Standard follow-up — Patients enrolled into standard group will be followed in a standard way without any additional procedure except randomization that allocates to the standard group
  Arms: Without learning workshops
Other: Learning workshops — Patients enrolled into experimental arm will participate to educative workshops before and after surgery for breast cancer. The aim of these workshop is to educate patient to self massages and self stretching.
  Arms: With learning workshops

SUMMARY:
Myofascial pain syndrome is a common cause of chronic pain characterized by myofascial pain and trigger points. Recommendations regarding management of pain after breast cancer don't mention myofascial syndrome despite a study suggests possible myofascial syndrome with roughly 75% of patients in pain.

144 patients having a local breast cancer requiring surgery will be randomized in this study, ratio 1:1 standard and experimental groups.

Every patients (standard and experimental groups) will attend 4 specific consultations during which standard recommendations will be given, pain, quality of life, shoulder range of motion, global upper limbs force will be assessed.

In addition, patient randomized in experimental group will attend self massages and self stretching workshops, one before surgery and one after surgery. Patients will be encouraged to performed daily self massages and self stretching.

The aim of the study is to assess impact of self massages and self stretching workshops on sequelae pain further surgery for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Woman
* Local development of breast cancer, every stages except stage IV
* Indication of surgery whatever surgery type except breast reconstruction
* More than18 years
* Life expectancy > 12 months assessed by surgeon or pain specialist
* Informed and written consent
* Affiliated to a social security system

Exclusion Criteria:

* History of chronic pain
* History of shoulder pain
* Any illness or severe disease, medical or psychiatric, that could prevent the patient to follow study procedures or to give her informed consent, according investigators,
* History of breast surgery
* Pregnant or lactating woman
* Protected adult or deprived of her liberty

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Impact of Learning workshops (self massages and self stretching) on sequelae pain after breast cancer surgery | For 12 months after surgery
  Number of patients with chronic pain

SECONDARY OUTCOMES:
Impact of patient quality of life | at 3, 6 and 12 months
  Assessed by EORTC Quality of Life Questionnaire Core questionnaire 30 scale

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie THEBAULT, Principal Investigator — Centre Eugène Marquis
Locations (1):
- Centre Eugène Marquis, Rennes, France

IPD SHARING:
Plan to Share IPD: No